CLINICAL TRIAL: NCT04343196
Title: Application of Digital Variance Angiography in Diagnostic Lower Limb Angiographiy for Radiation Exposure Reduction a Prospective Randomized Clinical Trial
Brief Title: Digital Variance Angiography in Diagnostic Angiographies for Effective Radiation Dose Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinepict Health Ltd. (Network)
Collaborators: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Kinepict-008
Record Dates: First submitted 2020-04-06; First posted 2020-04-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease; Femoral Artery Stenosis; Femoral Artery Occlusion; Popliteal Stenosis; Iliac Artery Stenosis; Crural Artery Thrombosis; Limb Ischemia
Keywords: Radiation protection; X-ray angiography; Digital Variance Angiography; Digital Subtraction Angiography; Peripheral Arterial Disease; Kinepict; Image acquistion; Image quality; Radiation exposure
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: All enrolled participants will undergo a diagnostic lower limb angiography, but the image acquisition protocol will be different. In the active comparator group a normal radiation dose will be used and the DSA images will be used for diagnosis whereas in the experimental group a low dose radiation will be applied (70% decrease compared tot he DSA protocol) and the DVA images will be used for diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Low-dose DVA group (Experimental): Image acquisition at a reduced X-ray dose, 0.36 µGy/frame (70% reduction) image processing by DVA
  Interventions: Radiation: Diagnostic Angiography (DSA or DVA based on randomization result)
- Group B: Normal-dose DSA group (Active Comparator): Image acquisition at a normal dose (1.2 µGy/frame) image processing by DSA
  Interventions: Radiation: Diagnostic Angiography (DSA or DVA based on randomization result)

INTERVENTIONS:
Radiation: Diagnostic Angiography (DSA or DVA based on randomization result) — After radial/brachial/femoral artery puncture using Seldinger technique, the investigators first position a pigtail catheter above the level of the renal arteries. With Siemens Artis Zee Pure DSA machine the examiner will use a postero-anterior X-ray view for the first image, which is an aortography of some part of the iliac system. Then, the catheter will be repositioned to the aortic bifurcation and 15-18 mL contrast media (CM) with 9-10 mL/s flow for the ilio-femoral region will be injected. All of the following image series will be made from this catheter position, with a 9 mL/s flow rate. In cases for when the recorded image series will be inconclusive, image series with left/right oblique position will be recorded. All femoro-popliteal images will be recorded with 10-16 ml CM and crural regions with 12-22mml. DSA images will be calculated from all series on a dedicated Syngo workstation and used for diagnosis. DVA images will be calculated by the Kinepict Medical Imaging Tool

SUMMARY:
Digital Variance Angiography (DVA) is a new tool in medical imaging with proven image quality reserve.

The previously observed quality reserve of Digital Variance Angiography (DVA) in lower extremity angiographies, allowed to lower radiation exposure by 70 % during DSA in lower extremity diagnostic angiographies with non-inferior image quality.

The aim of this study is to apply this non-inferior image quality and use it for radiation exposure reduction in diagnostic lower limb angiography.

The project would prospectively block-randomise (50:50) patients, who undergo elective diagnostic angiography into two groups: a comparator group examined by means of conventional DSA using a standard care protocol (Siemens Artis Zee, Extremities Care setting, 1.2 µGy/frame) (Group B) and a study group examined by means of DVA using a low-dose protocol (0.36 µGy/frame corresponding to 70% decrease of radiation dose) (Group A). During each procedure the investigators record radiation exposure (cumulative dosage, dose area product) and contrast media usage and procedural time then compare the results of the groups. Qualitative image review is done to compare conventional DSA and reduced radiation exposure DVA images after image acquisition.

Our hypothesis is that with the previously proven non-inferior image quality, the investigators will be able to reduce radiation exposure of the participants and also staff members in everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower limb peripheral arterial disease, admitted for diagnostic angiography
* Fontaine II- IV
* Normal renal function: GFR> 60ml/min/m2
* Age > 18

Exclusion Criteria:

* Acute myocardial infarction
* Severe heart/liver/renal failure
* Iodine contrast allergy
* Atrioventricular block
* Coagulopathy and Hematological Bleeding Disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Total procedural Dose-area product(DAP) | During the procedure
  Indicator of a patient's irradiation dosage (microGy*cm2 or Gy*cm2)
Total DSA-related DAP | During the procedure
  Radiation load of the patient during DSA image acquistion (microGy*cm2 or Gy*cm2)
Image quality review | Upon completion of enrollment, approximately 1-year period
  Blinded, anonymised and randomised qualitative review and comparison of images by multiple endovascular specialists in multiple regions using a 1-5 Likert-scale for each image. Region specific scores are compared between DSA and DVA technique.
TASC classification | Upon completion of enrollment, approximately 1-year period
  Blinded, anonymised and randomised review of images by multiple endovascular specialists. Clinically relevant sides for each patient are reviewed in a separate questionnaire: each reviewer have to classify each patient's angiographic image according to the Trans-Atlantic Inter-Society Consensus Document's second version.

SECONDARY OUTCOMES:
Contrast media usage | During the procedure
  The volume of the iodinated contrast agent used for enhancing the image quality (mL)
Number of protocol change | During the procedure
  The number of occasions when the reduced radiation level protocol has to be switched back to conventional protocol in one region because of unsuitable image quality.
Procedure time | During the procedure
  Duration of the whole procedure, from radial artery puncture till the removal of every tool (min).

CONTACTS AND LOCATIONS:
Overall Officials: Krisztián Szigeti, Ph.D., Study Chair — Kinepict Health Ltd.; Szabolcs Osváth, Ph.D., Study Chair — Kinepict Health Ltd.; János Kiss, M.D.,Ph.D.,D.Sc., Study Chair — Kinepict Health Ltd.
Locations (1):
- Semmelweis University, Heart and Vascular Center, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orias VI, Gyano M, Gog I, Szollosi D, Veres DS, Nagy Z, Csobay-Novak C, Zoltan O, Kiss JP, Osvath S, Szigeti K, Zoltan R, Sotonyi P. Digital Variance Angiography as a Paradigm Shift in Carbon Dioxide Angiography. Invest Radiol. 2019 Jul;54(7):428-436. doi: 10.1097/RLI.0000000000000555. PMID 30829769
- [Background] Gyano M, Gog I, Orias VI, Ruzsa Z, Nemes B, Csobay-Novak C, Olah Z, Nagy Z, Merkely B, Szigeti K, Osvath S, Sotonyi P. Kinetic Imaging in Lower Extremity Arteriography: Comparison to Digital Subtraction Angiography. Radiology. 2019 Jan;290(1):246-253. doi: 10.1148/radiol.2018172927. Epub 2018 Oct 16. PMID 30325284
- See also: Homepage for the Kinepict scientific group, source for additional information about digital variance angiography — http://kinepict.com